CLINICAL TRIAL: NCT04430569
Title: A Reduced Dose of Thrombolytic Treatment for Patients With Intermediate High-risk Acute Pulmonary Embolism: a Randomized Controled Trial
Brief Title: Pulmonary Embolism International THrOmbolysis Study-3
Acronym: PEITHO-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Life Sciences Research Partners (D Collen Research Foundation) (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Instituto de Salud Carlos III (Other Government); International Network of VENous Thromboembolism Clinical Research Networks (Unknown); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P160924; P160924 (Other: Assistance Publique - Hôpitaux de Paris); PHRCN-16-0580 (Other Grant/Funding Number: French ministry of Health); 2018-000816-96 (EudraCT Number)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism
Keywords: Intermediate-high-risk acute pulmonary embolism; Thrombolysis
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alteplase (Experimental)
  Interventions: Drug: Alteplase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alteplase — Alteplase single intravenous infusion of 0.6 mg/kg of estimated bodyweight with a maximum of 50 mg given over 15 minutes.
  Arms: Alteplase
Drug: Placebo — Placebo single intravenous infusion of 0.6 mg/kg of estimated bodyweight with a maximum of 50 mg given over 15 minutes.
  Arms: Placebo

SUMMARY:
In this study, we will assess the efficacy and safety of a reduced dose of thrombolytic therapy given in addition to low-molecular-weight heparin in patients with intermediate-high-risk acute pulmonary embolism. Half of participants will receive thrombolytic treatment, while the other half will receive a placebo.

DETAILED DESCRIPTION:
In patients with intermediate-risk pulmonary embolism, full-dose thrombolytic treatment was associated with a reduction in the combined risk of hemodynamic instability or death but was also associated with an increased risk of major and intracranial bleeding. Previous studies suggest that reduced dose of thrombolytic treatment may be as effective as the full dosage, but with a decreased risk of life-threatening bleeding. In this study, we will assess the efficacy and safety of a reduced dosage of thrombolytic therapy in patients with intermediate-high-risk acute pulmonary embolism.

The study is a randomized, placebo-controlled, double blind, multicenter, multinational trial with long-term follow-up.

Patients fulfilling the inclusion criteria and without any of the exclusion criteria will be randomized within 6 hours after the investigator had confirmed the diagnosis.

Patients will receive:

* Alteplase (if randomized in the experimental group) or placebo (if randomized in the reference group) given within 30 minutes of randomization as a 15 min intravenous infusion at a dosage of 0.6 mg/kg with a total dose not exceeding 50 mg.
* Parenteral anticoagulation with low molecular weight heparin, unfractionnated heparin or fondaparinux

Primary objective is to assess the efficacy of reduced dose thrombolytic therapy in patients with acute intermediate-high-risk pulmonary embolism at day 30.

Secondary objectives are:

1. To assess the safety of reduced dose thrombolytic therapy in patients with intermediate-high-risk acute pulmonary embolism at day 30
2. To assess the net clinical benefit of reduced dose thrombolytic therapy in patients with intermediate-high-risk acute pulmonary embolism at day 30
3. To assess the effect of reduced dose thrombolytic therapy on overall mortality of patients with intermediate-high-risk acute pulmonary embolism at day 30
4. To assess the effect of reduced dose thrombolytic therapy on long-term mortality, functional impairment, residual right ventricular dysfunction and chronic thromboembolic pulmonary hypertension at 6 months and 2 years
5. To assess the effect of reduced-dose thrombolytic therapy on utilization of health care resources at day 30 and day 180

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Objectively confirmed acute PE with first symptoms occurring 2 weeks or less before randomization. Objective confirmation is based on at least one of the following criteria: (a) at least one segmental ventilation-perfusion mismatch on lung scanning; (b) a spiral computed tomography pulmonary angiography or pulmonary angiography showing a filling defect or an abrupt obstruction of a segmental or more proximal pulmonary artery
* Acute PE confirmed within 24 hours prior to randomization
* Elevated risk of early death, or of hemodynamic collapse, or PE recurrence, indicated by at least one of the following criteria: (a) systolic blood pressure ≤ 110 mm Hg over at least 15 minutes upon enrolment, (b) temporary need for fluid resuscitation and/or treatment with low-dose catecholamines, provided that the patient could be stabilized within 2 hours of admission and maintains SBP of ≥ 90 mmHg and adequate organ perfusion without catecholamine infusion; (c) respiratory rate > 20/min or oxygen saturation on pulse oximetry SpO2 <90% o(or partial arterial oxygen pressure < 60 mm Hg) at rest while breathing room air, (d) documented history of chronic symptomatic heart failure
* Right ventricular dysfunction indicated by RV/LV diameter ratio >1.0 on echocardiography apical four-chamber or subcostal four-chamber view or on Computed Tomography Pulmonary Angiography (transverse plane)
* Serum troponin I or T concentration above the upper limit of local normal using a high-sensitivity assay
* Ability to randomize the patient within 6 hours after the investigator receives the results of the second of the two criteria for RV dysfunction (RV/LV diameter ratio >1.0) and myocardial injury (serum troponin I or T concentration above the upper limit of local normal), whichever comes latest.
* Signed informed consent form

Exclusion Criteria:

* Hemodynamic instability
* Active bleeding
* History of non-traumatic intracranial bleeding, any time
* Acute ischemic stroke or transient ischemic attack (TIA) within the previous 6 months
* Known central nervous system neoplasm/metastasis
* Neurologic, ophthalmologic, abdominal, cardiac, thoracic, vascular or orthopedic surgery or trauma within 3 previous weeks
* Platelet count < 100 G/L
* INR > 1.4. If INR not available: prothrombin time ratio < 60%. If both INR and prothrombin time ratio are measured, INR is relevant for the assessment of this criterion.
* Treatment with antiplatelet agents other than (a) acetylsalicylic acid (ASA) ≤ 100 mg once daily or (b) clopidogrel 75 mg once daily or (c) a single loading dose of ASA or clopidogrel. Dual antiplatelet therapy (ASA + clopidogrel) is not allowed.
* Any direct oral anticoagulant within 12 hours of inclusion
* Uncontrolled hypertension defined by SBP > 180 mm Hg at the time of inclusion
* Known pericarditis or endocarditis
* Known significant bleeding risk according to the investigator's judgement
* Administration of thrombolytic agents within the previous 4 days
* Vena cava filter insertion or pulmonary thrombectomy within the previous 4 days
* Current participation in another interventional clinical study
* Previous enrolment in this study
* Known hypersensitivity to alteplase, gentamicin (a residue of the Actilyse® manufacturing process present in trace amounts), any of the excipients of Actilyse®, or low-molecular weight heparin (LMWH)
* Known previous immune heparin-induced thrombocytopenia
* Known severe liver disease (grade ≥ 3) including liver failure, cirrhosis, portal hypertension (esophageal varices) and active hepatitis
* Acute symptomatic pancreatitis
* Gastrointestinal ulcers or esophageal varices, documented within the past 3 months
* Known arterial aneurysm, arterial or venous malformations
* Pregnancy or parturition within the previous 30 days or current breastfeeding.
* Women of childbearing potential who do not have a negative pregnancy test at the inclusion visit and do not use one of the following methods of birth control: hormonal contraception or intrauterine device or bilateral tubal occlusion
* Any other condition that the investigator feels would place the patient at increased risk upon start of the investigational treatment
* Life expectancy of less than 6 months or inability to complete 6-month follow-up.
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Composite of (1) death from any cause or (2) hemodynamic decompensation or (3) objectively confirmed recurrent PE. | 30 days

SECONDARY OUTCOMES:
Fatal or GUSTO severe or life threatening bleeding | 30 days
Composite of the primary efficacy endpoint and GUSTO severe or life-threatening bleeding | 30 days
  Assessment of net clinical benefit
All-cause mortality | 30 days
PE related death | 30 days
Hemodynamic decompensation | 30 days
Recurrent PE | 30 days
Need for rescue thrombolysis, catheter-directed treatment or surgical embolectomy | 30 days
Ischemic or hemorrhagic stroke | 30 days
Serious adverse events | 30 days
Persisting dyspnea | 180 days
Persisting dyspnea | 2 years
Persistent right ventricular dysfunction | 180 days
Persistent right ventricular dysfunction | 2 years
Functional outcome | 180 days
Functional outcome | 2 years
All-cause mortality | 2 years
Confirmed chronic thromboembolic pulmonary hypertension | 2 years
Utilization of health care ressources | 30 days
  Questionnaire assessing the impact of the treatment on utilization of health care ressources
Utilization of health care ressources | 180 days
  Questionnaire assessing the impact of the treatment on utilization of health care ressources

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SANCHEZ, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Stavros Konstantinides, MD, Principal Investigator — University Medical Center Mainz
Locations (97):
- Austria (2):
  - Graz, Mediz Universität, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
- Belgium (3):
  - UCL Brussels, Brussels
  - KU Leuven, Leuven
  - CHU Liège, Liège
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - Juravinski Hospital - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Hamilton General Hospital - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hopsital, General and Civic campuses, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (22):
  - CHU d'Angers, Angers
  - CHU de Besançon - Hôpital Jean-Minjoz, Besançon
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest
  - CHU de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU de Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - AP-HP - hôpital Henri-Mondor, Créteil
  - CHU de Grenoble - Hôpital Michallon, La Tronche
  - AP-HP - hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lille - Institut Cœur Poumon, Lille
  - HCL - Hôpital Edouard Herriot, Lyon
  - HCL - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Lyon
  - AP-HM - Hôpital de la Timone, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nice - Hôpital Pasteur, Nice
  - AP-HP - Hôpital Lariboisière, Paris
  - AP-HP - hôpital européen Georges-Pompidou, Paris
  - AP-HP - Hôpital Bichat-Claude-Bernard, Paris
  - AP-HP - Hôpital Tenon, Paris
  - HCL - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Saint-Étienne - Hôpital Nord, Saint-Etienne
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
- Germany (17):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - DRK Kliniken Berlin Köpenick, Berlin
  - Berlin, DRK Kliniken Westend, Berlin
  - Augustinerinnen Hospital, Cologne
  - Cologne Universität Herzzentrum, Cologne
  - Dresden, Städtisches Klinikum, Dresden
  - Düsseldorf, Augusta-Krankenhaus, Düsseldorf
  - Freiburg Universität, Freiburg im Breisgau
  - Greifswald, Univ.-Medizin, Greifswald
  - Hannover, Medizinische Hochschule Hannover, Hanover
  - Leipzig, Univ.-Klinikum, Leipzig
  - Mainz Universitätsmedizin, CTH, Mainz
  - Mainz, Katholisches Klinikum, Mainz
  - Universitätsmedizin Mannheim UMM, Mannheim
  - Regensburg, Uniklinik, Regensburg
  - Tübingen, Univ.-Klinikum, Tübingen
  - Ulm, Universitätsklinikum, Ulm
- Italy (7):
  - University Hospital Ancona / Ospedali Riunit, Ancona
  - Spedali Riuniti - Cremona, Cremona
  - Ospedale San Giuseppe - Empoli, Empoli
  - Azienda Ospedaliera Careggi - Firenze, Florence
  - Humanitas Hospital - Milano, Milan
  - University of Perugia, Perugia
  - Ospedale Ca Foncello - Treviso, Treviso
- Netherlands (7):
  - Catharina hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Martini hospital, Groningen
  - Maasstad hospital, Rotterdam
  - Antonius hospital, Sneek
  - Haaglanden hospital, The Hague
  - Isala hospital, Zwolle
- Poland (6):
  - Medical University of Bialystok, Bialystok
  - Department of Cardiac and Vascular Diseases, Krakow
  - Medical University of Lodz, Lodz
  - University of Warmia Mazury in Olsztyn - School of Medicine, Olsztyn
  - Poznan University of Medical Sciences, Poznan
  - Medical University of Warsaw, Warsaw
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar de Lisboa Norte/ Hospitalde Santa Maria, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar de Setubal, Setúbal
- Romania (5):
  - Spitalul Judetean de Urgenta Baia Mare, Baia Mare
  - Bucuresti - Spitalul Clinic de Urgenta Sf. Pantelimon, Bucharest
  - Spitalul Judetean de Urgenta Constanta, Constanța
  - Iasi - St Spiridon Emergency Conty Hospital, Iași
  - Institutul de Boli Cardio-Vasculare Timisoara, Timișoara
- Serbia (3):
  - Cardiology Clinic, Emergency Center, Clinical Center of Serbia, Belgrade
  - Cardiology Clinic, Clinical Center of Niš, Niš
  - Institute for Lung Diseases of Vojvodina, Sremska Kamenica, Novi Sad
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (9):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital Bellvitge, Barcelona
  - Hospital Cartagena, Cartagena
  - Hospital Galdakao, Galdakao
  - Clínica Universitaria Navarra, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital La Fe, Valencia
- Switzerland (2):
  - Geneva University Hospital, Geneva
  - Hôpital du Valais, Sion

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.

REFERENCES:
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Barco S, Vicaut E, Klok FA, Lankeit M, Meyer G, Konstantinides SV; PEITHO Investigators. Improved identification of thrombolysis candidates amongst intermediate-risk pulmonary embolism patients: implications for future trials. Eur Respir J. 2018 Jan 18;51(1):1701775. doi: 10.1183/13993003.01775-2017. Print 2018 Jan. No abstract available. PMID 29348184
- [Background] Konstantinides SV, Vicaut E, Danays T, Becattini C, Bertoletti L, Beyer-Westendorf J, Bouvaist H, Couturaud F, Dellas C, Duerschmied D, Empen K, Ferrari E, Galie N, Jimenez D, Kostrubiec M, Kozak M, Kupatt C, Lang IM, Lankeit M, Meneveau N, Palazzini M, Pruszczyk P, Rugolotto M, Salvi A, Sanchez O, Schellong S, Sobkowicz B, Meyer G. Impact of Thrombolytic Therapy on the Long-Term Outcome of Intermediate-Risk Pulmonary Embolism. J Am Coll Cardiol. 2017 Mar 28;69(12):1536-1544. doi: 10.1016/j.jacc.2016.12.039. PMID 28335835
- [Background] Marti C, John G, Konstantinides S, Combescure C, Sanchez O, Lankeit M, Meyer G, Perrier A. Systemic thrombolytic therapy for acute pulmonary embolism: a systematic review and meta-analysis. Eur Heart J. 2015 Mar 7;36(10):605-14. doi: 10.1093/eurheartj/ehu218. Epub 2014 Jun 10. PMID 24917641
- [Background] Sanchez O, Charles-Nelson A, Ageno W, Barco S, Binder H, Chatellier G, Duerschmied D, Empen K, Ferreira M, Girard P, Huisman MV, Jimenez D, Katsahian S, Kozak M, Lankeit M, Meneveau N, Pruszczyk P, Petris A, Righini M, Rosenkranz S, Schellong S, Stefanovic B, Verhamme P, de Wit K, Vicaut E, Zirlik A, Konstantinides SV, Meyer G; PEITHO-3 Investigators. Reduced-Dose Intravenous Thrombolysis for Acute Intermediate-High-risk Pulmonary Embolism: Rationale and Design of the Pulmonary Embolism International THrOmbolysis (PEITHO)-3 trial. Thromb Haemost. 2022 May;122(5):857-866. doi: 10.1055/a-1653-4699. Epub 2021 Oct 31. PMID 34560806